CLINICAL TRIAL: NCT06563427
Title: A Multicenter Study on the Reliability of Four Ultrasound Measures : the Antero-posterior Diameter , the End-exipratory Area , the Aspect Ratio and the Collapsibility Index of Internal Jugular Vein Evaluated on Patients Admitted to Five Medicine Departments
Brief Title: Reliability of Internal Jugular Ultrasound : an Observational Transversal Study (AIJV)
Acronym: AIJV
Status: Completed | Type: Observational
Sponsor: Maggiore Bellaria Hospital, Bologna (Other)
Responsible Party: Principal Investigator, Nicola Parenti, MD, Maggiore Bellaria Hospital, Bologna
Other Study IDs: 725-2023-OSS-AUSLBO
Record Dates: First submitted 2024-08-19; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Diagnosis; Vascular Diseases
Keywords: ultrasound; reliability; jugular vein
MeSH Terms: conditions — Disease; Vascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational transversal study without intervention on the inter-rater reliability of four ultrasound measures of Internal Jugular Veins.

Aims are : 1) to test the inter-rater reliability among a group of ultrasound measurements of internal jugular vein using a group of images, registered in several acoustic views of neck of patients admitted in Internal Medicine Dept of five Italian Hospitals ; 2)to measure the differences between ultrasound measurements in different acoustic views .

The reliability will be tested by recording Ultrasound measures on images registered using an Utrasound protocol on 100 patients.

DETAILED DESCRIPTION:
Introduction Many studies suggest that the ultrasound of Internal Jugular Vein (IJV) is a method valid in predicting volume status and Central Venous Pressure (CVP) among critical patients (1-2).

Because this method is very easy , fast and applicable in several setting , if research will confirm its accuracy in detecting congestion and prognosis , it could have an important role in clinical practice.

The Internal jugular vein changes its size during the respiratory cicle : it enlarges in expiration and reduces in inspiration .

Usually the expiratory (maximum) diameters and area have been used by researchers to test the IJV ultrasound accuracy in predicting Central Venous Pressure and volume status (1,2).

Many ultrasound measures of IJV have been tested (3-8 ) : the antero-posterior , end-expiratory Internal Jugular Vein diameter (AP-IJV max); the end-exipratory IJV area (maximal area in transversal section, CSA-IJV max) ; the ratio between the AP-IJV max and transversal IJV diameter (LL-IJV max) , the Aspect ratio= AP-IJV max/LL-IJV max; the Collapsibility index of IJV , the respiratory variation percentage calculated as [(maximum diameter minus minimum diameter)/maximum diameter].

According to the literature, a low value of the collapsibility index suggests high Central Venous Pressure (CVP). Large diameters and areas of the internal jugular vein are recorded in patients with high CVP.

Unfortunately, many factors could affect IJV measurements using Ultrasound: patient position, the side of exam (right vs left ), previous neck surgery, IJV thrombosis, presence of catheters .

Furthermore, there is not a standardization of ultrasound technique because the researchers used several protocols to validate the method .

For these reasons our hypothesis is that the IJV ultrasound might have a great inter-rater variability and that it is not reliable .

Therefore our aim is to test the inter-rater reliability among a group of ultrasound measurements of internal jugular vein using a group of images, registered in several acoustic views of neck of patients admitted in Internal Medicine Dept of five Italian Hospitals .

Secondary objective is: to measure the differences between ultrasound measurements in different acoustic views .

Methods Design , setting and data collection It's a cross-sectional transversal observational study, that will be conducted in five Italian Hospitals from September 1 , 2024 to September 30, 2024. We will follow the Strobe checklist and guidelines to plan and conduct the study (9).

The study has been approved by the Ethical Committee Area Vasta Emilia Centro (AVEC) , code : 725-2023-OSS-AUSLBO.

For each patient the following variables will be collected: age, sex, weight, height, Body mass index, Body surface area, cause of hospitalization and ultrasound measurements of the jugular below described.

Ultrasound imaging and protocol During the ultrasound examination, that will be performed using an Esaote Mylab system, the patients will be with the trunk at 45 °. The examination will be performed in the lateral region of the right neck, using the following acoustic windows: supraclavicular ( two cm above the clavicle), cricoid and at the apex of the sternocleidomastoid muscle (mandibular angle).

A vascular probe (10 Mhz linear array) will be used in B Mode and M Mode . Six images per patient will be recorded by the twenty patients recruited, for a total of 120 images.

The sonographers, after a short theoretical and practical course (one hour of theory and one hour of practice ), will measure , on the images previously recorded , independently and without communicating with each other , the four ultrasound measurements to be tested, illustrated in the Figure 1-4 of the Appendix : the Antero-posterior expiratory max diameter ( AP-IJV max), maximum area ( CSA-IJV max), the Aspect ratio (AP-IJV max / Ll-IJV), the collapsibility index ( IJV-c).

To avoid bias of selection of participants, all patients , admitted to each cause in the Study Center, will be recruited. The ultrasound researchers will not know the purpose of the study , the causes of hospitalization of the patient nor the values of measurements made by the other researchers-echographers. The researcher who will collect the clinical-anagraphic data and the ultrasound variables will be not the same researcher who will performe the ultrasound protocol.

To avoid the biases of procedure and measurement of ultrasound variables, sonograpfers who will perform the protocol will be instructed , before the study, with the same course, conducted by the same teacher.

Each researcher will not know the measurements recorded by the other researchers in the same session.

To calculate the sample estimate , we predict an expected value of ICC=0.9; a minimum acceptable value of ICC=0.6 , according to the literature (3, 10 ); a statistical significance level of 0.05 (alpha error); a rater number of 12 (11 students and the "gold standard") ; a 10% share of lost data.

In this way, using the calculation method described in the link https:///wnarifin.github.io/ssc/ssicc.html, we estimate that a sample of 10 groups of images would be needed for global reliability.

The medians and relative Interquartile (IQR) ranges of the ultrasound measurements will be compared in the different acoustic windows.

Reliability values, measured with the ICC (inter-class correlation coefficient), among the sonographers of the 5 hospitals will be also compared.

Statistical analysis The median and range Interquartile (IQR) and , Box plot will be used to describe and present the collected data . We consider statistically significant a value of p less than 0.05.

To evaluate inter-operator reliability, ICC (inter-class correlation coefficient) statistics will be used, a measure that has a range of values between zero, expression of maximum variability and the one , high reliability and minimum variability.

We use the reliability level classification proposed by Koo TK et al (11): we consider poor realiability an ICC value less than 0.5 ; moderate an ICC value = 0.5-0.75; good an ICC= 0.75-0.9; an excellent ICC=0.9.

References

1. Wang MK , Piticaru J , Kappe C · Mikhaeil M , Mbuagbaw L Internal jugular vein ultrasound for the diagnosis of hypovolemia and hypervolemia in acutely ill adults: a systematic review and meta analysis Internal and Emergency Medicine (2022) 17:1521-1532 .
2. Parenti N et al Role of Internal Jugular Vein Ultrasound Measurements in the Assessment of Central Venous Pressure in Spontaneously Breathing Patients: A Systematic Review Journal of Acute Medicine 9(2): 39-48, 2019
3. Simon MA, Kliner DE, Girod JP, Moguillansky D, Villanueva F et al Detection of elevated right atrial pressure using a simple bedside ultrasound measure Am Heart J 2010;159:421-7.
4. Simon MA , Schnatz RG, Jared D. Romeo JD, Pacella JJ Bedside Ultrasound Assessment of Jugular Venous Compliance as a Potential Point-of-Care Method to Predict Acute Decompensated Heart Failure 30-Day Readmission J Am Heart Assoc. 2018 Aug 7;7(15)
5. Tzadok B, Shapira S, Tal-Or E Ultrasound of Jugular Veins for Assessment of Acute Dyspnea in Emergency Departments and for the Assessment of Acute Heart Failure Isr Med Assoc J . 2018 May;20(5):308-310.
6. Vaidya GN , Ghafghazi S Correlation of internal jugular and subclavian vein diameter variation on bedside ultrasound with invasive right heart catheterization Indian Heart J . Mar-Apr 2021;73(2):231-235.
7. Ammirati E, Marchetti D, Colombo G, Pellicori P, Gentile P , D'Angelo L et al Estimation of Right Atrial Pressure by Ultrasound-Assessed Jugular Vein Distensibility in Patients With Heart Failure. Circ Heart Fail . 2024 Feb;17(2):e010973. doi: 10.1161/CIRCHEARTFAILURE.123.010973. Epub 2024 Feb 1.
8. Albaeni A, Sharma M, Ahmad M, Khalife WI Accurate Estimation of Right-Filling Pressure Using Handheld Ultrasound Score in Patients with Heart Failure Am J Med . 2022 May;135(5):634-640. doi: 10.1016/j.amjmed.2021.11.020. Epub 2021 Dec 31.
9. Von Elm E, Altman DG, Egger M, Pocock SJ, Gøtzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE)statement: guidelines for reporting observational studies. J Clin Epidemiol. 2008 Apr;61(4):344-9. PMID: 18313558
10. Donahue SP, Wood JP, Patel BM, Quinn JV. Correlation of sonographic measurements of the internal jugular vein with central venous pressure. Am J Emerg Med 2009;27:851-855. doi:10.1016/j.ajem.2008.06.005
11. Koo TK, Li MY A Guideline of Selecting and Reporting Intraclass Correlation Coefficients for Reliability Research J Chiropr Med . 2016 Jun;15(2):155-63. doi: 10.1016/j.jcm.2016.02.012

ELIGIBILITY:
Inclusion Criteria:

Twenty adult patients, admitted to four Internal Medicine Departments and one Vascular Surgery Clinic; ten sonographers with Ultrasound Certification.

Exclusion Criteria:

impossibility in providing consent, presence of central venous catheter in the internal jugular vein, thrombosis of the vein.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to each cause in the Study Center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
inter-rater reliability | From 1st march 2024 to 30th July 2024
  the variability in the recording of ultrasound measurements among sonographers from differente centers

SECONDARY OUTCOMES:
statistical significance of differences of ultarsound measurements | From 1st march 2024 to 30th July 2024
  differences of ultrasound measurements among different acoustic views

CONTACTS AND LOCATIONS:
Overall Officials: AUSL Bologna, Study Chair — Maggiore Hospital
Locations (1):
- Nicola Parenti, Bologna, Italy